CLINICAL TRIAL: NCT00002485
Title: Barriers to Patient Enrollment Onto Frontline Therapeutic Clinical Trials and Development of Intervention Strategies to Increase the Proportion of Enrollment
Brief Title: Development of Strategies to Increase Enrollment in Clinical Trials for Children With Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9284; POG-9284/9285 (Other: Pediatric Oncology Group); NCI-P92-0003; CDR0000077305 (Other: Clinicaltrials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-04-26 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Leukemia; Liver Cancer; Lymphoma; Neuroblastoma; Ovarian Cancer; Psychosocial Effects of Cancer and Its Treatment; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: localized osteosarcoma; metastatic osteosarcoma; recurrent childhood acute lymphoblastic leukemia; childhood infratentorial ependymoma; childhood low-grade cerebral astrocytoma; childhood supratentorial ependymoma; childhood craniopharyngioma; localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; stage I childhood liver cancer; stage II childhood liver cancer; stage III childhood liver cancer; stage IV childhood liver cancer; recurrent childhood liver cancer; childhood hepatoblastoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; childhood central nervous system germ cell tumor; recurrent childhood acute myeloid leukemia; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific; childhood germ cell tumor; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; nonmetastatic childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; extragonadal germ cell tumor; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood meningioma; localized unresectable neuroblastoma; psychosocial effects of cancer and its treatment; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; untreated childhood supratentorial primitive neuroectodermal tumor; recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood medulloblastoma; recurrent childhood medulloblastoma; untreated childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway and hypothalamic glioma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Liver Neoplasms; Lymphoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Osteosarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hepatoblastoma; Recurrence; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms; Meningioma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma; Familial ependymoma; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer; Rhabdoid Tumor | interventions — Psychiatric Rehabilitation

GROUPS / COHORTS (2):
- Stratum 1: Not Enrolled / No IRB Applied
  Interventions: Procedure: psychosocial assessment and care
- Stratum 2: Not Enrolled / IRB Approved
  Interventions: Procedure: psychosocial assessment and care

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Taking part in a clinical trial may help children with cancer receive more effective treatment.

PURPOSE: Determine why patients who are eligible for protocols made available through the Pediatric Oncology Group do not enroll in them, and develop strategies to increase enrollment on these clinical trials.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify prospectively physician and patient factors associated with reasons why patients who are eligible for Pediatric Oncology Group therapeutic protocols are not enrolled onto such studies. II. Provide information that may be used to develop intervention strategies to decrease barriers to patient enrollment, thus increasing enrollment in therapeutic protocols.

OUTLINE: This is a case-control, multicenter study. Case patients are stratified. Stratum 1 comprises patients for whom there is an appropriate Pediatric Oncology Group (POG) frontline therapeutic protocol that has not yet been submitted to, disapproved by, or approved by the Institutional Review Board (IRB). Stratum 2 comprises patients for whom there is an appropriate POG frontline therapeutic protocol that has been approved by the IRB. Physicians complete an IRB submission form for their patients on stratum 1. Patients/parents on stratum 2 who refused enrollment and their primary physicians complete questionnaires that address reasons for nonenrollment. Control patients/parents who consented to enrollment complete questionnaires that address reasons for enrollment. Demographic information, including the size of the treating institution and the annual number of patients enrolled onto its protocols, is collected. Additional demographic information regarding the patient and his or her family is collected.

PROJECTED ACCRUAL: A total of 595 case patients (12 with soft tissue sarcoma, 34 with osteosarcoma, 19 with brain tumors, 32 with Hodgkin's disease, 60 with non-Hodgkin's lymphoma, 278 with acute lymphoblastic leukemia, 65 with acute non-lymphoblastic leukemia, 56 with neuroblastoma, 14 with hepatoblastoma, and 25 with germ cell tumors) will be accrued for this study within 7 years. Corresponding control patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Case or control patient clinically eligible for a Pediatric Oncology Group (POG) frontline therapeutic protocol, whether or not the protocol was submitted to or approved by the physician's Institutional Review Board Case patients must not have enrolled on the POG frontline protocol due to decision by the physician or patient/parent Control patients must have been enrolled on the POG frontline protocol Ineligible if offered treatment on an in-house therapeutic protocol (institutional review board-approved) rather than the POG protocol

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 359 (Actual)
Dates: Start 1992-02; Primary Completion 2003-07 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Determine why eligible patients are not enrolled on available Pediatric Oncology Group therapeutic clinical trials.
  The variables of interest are those factors that affect the decision by the treating physician or patient/parent to refuse enrollment onto study.
  Physician responses and patient/parent responses as to reasons for non-enrollment will be compared. Analyses will assess patient demographic factors and institutional characteristics (including the size of the treating institution in terms of the number of patients enrolled on protocols annually). Additionally, reasons for non-enrollment will be assessed with regard to the size of the institution's cancer care program.

CONTACTS AND LOCATIONS:
Overall Officials: Brad H. Pollock, PhD, Study Chair — Pediatric Oncology Group Statistical Office
Locations (31):
- United States (26):
  - University of California Davis Medical Center, Sacramento, California
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Tomorrows Children's Institute, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - West Virginia University - Charleston Division, Charleston, West Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland